CLINICAL TRIAL: NCT01429389
Title: Collection of Whole Blood Specimens from Pregnant Women At Increased Risk of Fetal Chromosomal Abnormality for Use in Development of a Noninvasive Prenatal Test in the Detection of the Relative Quantity of Chromosomal Material in Circulating Cell-Free DNA Extracted from Maternal Plasma
Brief Title: Specimen Collection from Pregnant Women At Increased Risk for Fetal Aneuploidy
Status: Recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-107
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Down Syndrome; Fetal Aneuploidy
Keywords: Down syndrome; fetal aneuploidy; trisomy; noninvasive screening test
MeSH Terms: conditions — Down Syndrome; Trisomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens will be collected and processed to plasma. DNA will be extracted from the plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
The specimen collection is designed for the purpose of the development of a noninvasive prenatal test for T21.

DETAILED DESCRIPTION:
To collect specimens for the purpose of developing a prenatal aneuploidy test. The test will analyze circulating cell free fetal (ccff) nucleic acid from blood samples from pregnant women who have an increased risk indicator/s for fetal chromosomal aneuploidy and are undergoing invasive prenatal diagnosis by chorionic villus sampling (CVS) and/or genetic amniocentesis. The results of the ccff aneuploidy test will be compared to the chromosomal analysis obtained via CVS or genetic amniocentesis.

ELIGIBILITY:
Inclusion Criteria:

* pregnant between 10 and 22 weeks gestation
* 18 years of age or older
* provides signed and dated informed consent
* subject is at increased risk for fetal aneuploidy
* subject is willing to undergo a CVS and/or amniocentesis procedure for the purpose of genetic analysis
* subject agrees to provide the genetic results of the invasive procedure

Exclusion Criteria:

* Fetal demise at time of specimen sampling
* Previous sample donation under this protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women between 10 and 22 weeks of gestation who are scheduled to undergo a CVS or amniocentesis procedure and will receive the fetal FISH, karyotype and/or QF-PCR results from the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Grosu, MD, Study Director — Sequenom, Inc.
Locations (14):
- United States (12):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sharp-Rees Stealy Medical Group, San Diego, California
  - UCSD, San Diego, California
  - Women's Health Care Research, San Diego, California
  - Specialty Obstetrics of San Diego, San Diego, California
  - Reproductive Genetics Institute, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - The Cooper Health System, Camden, New Jersey
  - Medical University of South Carolina, Charleston, South Carolina
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Samples are used for research and development of a noninvasive prenatal test. However, samples used for publications will have data shared as defined by journal.